CLINICAL TRIAL: NCT02747472
Title: Involvement of Glucose-dependent Insulinotropic Polypeptide (GIP) in Human Physiology and Pathophysiology - Receptor Antagonist Studies in Humans
Brief Title: GIP Receptor Antagonist Studies in Humans
Acronym: GA-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Lærke Smidt Gasbjerg, MD, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: UHG-CFD-GIPANTA-1
Record Dates: First submitted 2016-04-19; First posted 2016-04-21 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Glucose Metabolism
Keywords: GIP; GIP receptor antagonist
MeSH Terms: interventions — gastric inhibitory polypeptide (1-42); Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator): Infusion of saline
  Interventions: Other: Saline
- GIP(1-42) (Active Comparator): Infusion of agonist, GIP(1-42)
  Interventions: Drug: GIP(1-42)
- GIP-A (Experimental): Infusion of GIP-A alone
  Interventions: Drug: GIP-A
- GIP-A + GIP(1-42) (Experimental): Infusion of GIP-A and GIP(1-42)
  Interventions: Drug: GIP-A; Drug: GIP(1-42)

INTERVENTIONS:
Drug: GIP-A — GIP receptor antagonist
  Arms: GIP-A; GIP-A + GIP(1-42)
Drug: GIP(1-42) — GIP receptor agonist
  Arms: GIP(1-42); GIP-A + GIP(1-42)
Other: Saline — Placebo
  Arms: Placebo

SUMMARY:
Antagonizing GIP effects during hyperglycaemia in healthy subjects and measurements of insulin secretion.

DETAILED DESCRIPTION:
Aim: To evaluate the GIP receptor antagonizing effect of peptide-based competitive GIP receptor antagonist GIP-A (vs. saline (placebo)) in 10 healthy subjects during 1 hour hyperglycaemic clamps with and without concomitant iv infusion of GIP[1-42]. The intention is to establish GIP-A as a tool to eliminate glucose-dependent insulinotropic GIP signalling.

The study consists of four experimental days (A-D) with assessment of beta cell function during 12 mM-hyperglycaemic clamps with concomitant infusions of A) GIP[1-42], B) GIP-A, C) GIP[1-42] + GIP-A, or D) saline (placebo).

ELIGIBILITY:
Inclusion Criteria:

* Normal kidney function, liver function and hemoglobin levels.

Exclusion Criteria:

* Medication, Diabetes type 1 or 2, BMI > 25, first degree relatives with Type 2 Diabetes

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2016-04; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Insulin levels | 65 minutes
  Serum-insulin AUC (area under the curve for hyperglycemic clamp period)

CONTACTS AND LOCATIONS:
Overall Officials: Filip K Knop, MD, PhD, Study Director — UHGentofte, Center for Diabetes Research
Locations (1):
- Center for Diabetes Research, Copenhagen, Gentofte, Denmark

REFERENCES:
- [Derived] Gasbjerg LS, Christensen MB, Hartmann B, Lanng AR, Sparre-Ulrich AH, Gabe MBN, Dela F, Vilsboll T, Holst JJ, Rosenkilde MM, Knop FK. GIP(3-30)NH2 is an efficacious GIP receptor antagonist in humans: a randomised, double-blinded, placebo-controlled, crossover study. Diabetologia. 2018 Feb;61(2):413-423. doi: 10.1007/s00125-017-4447-4. Epub 2017 Sep 25. PMID 28948296